CLINICAL TRIAL: NCT04905927
Title: Long Term Follow up of Failed Back Surgery Syndrome(FBSS) Patients With Korean Integrative Medicine Treatment: 10-year Follow-up Prospective Study With Survey
Brief Title: Long Term Follow up of Failed Back Surgery Syndrome(FBSS)
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2021-03
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Failed Back Surgery Syndrome; Integrative Medicine; Medicine, Korean Traditional
Keywords: integrative Korean medicine
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone survey — A questionnaire about the current symptoms and satisfaction for received treatment will be conducted over the phone for patients.

SUMMARY:
The purpose of this study is to reveal the effectiveness and satisfaction of integrative Korean medicine for Failed Back Surgery Syndrome(FBSS) by observation patients treated with integrative Korean medicine.

This study is a prospective observational study. The subjects for study are patients diagnosed with Failed Back Surgery Syndrome(FBSS) and who have been admitted to Gangnam Jaseng Hospital of Korean medicine and Bucheon Jaseng Hospital of Korean medicine for 2011.11-2014.09.

Medical records of selected patients will be analyzed, and telephone surveys will be conducted for each patient. The survey questions are Numeric rating scale (NRS), Oswestry disability index (ODI), quality of life, and Patient Global Impression of Change (PGIC), etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Failed Back Surgery Syndrome and was admitted to Jaseng hospital of Korean medicine.
* Patients have agreed to participate the study.
* Patients who had participated "Long-term course of failed back surgery syndrome (FBSS) patients receiving integrative Korean medicine treatment: a 1 year prospective observational multicenter study"
* Patients aged 19-70 years on the date

Exclusion Criteria:

* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects for study are patients diagnosed with Failed Back Surgery Syndrome and who have been admitted to two Jaseng Hospital of Korean medicine (Gangnam, Bucheon) for 2011.11-2014.09
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | Finish survey by June 2021
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS was assessed at admission, 2 weeks after admission, discharge, and long term follow up.

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | Finish survey by June 2021
  The ODI is a 10-item questionnaire developed to evaluate the degree of disability for low back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean ODI questionnaire
Korean-Short Form Healthy Survey 36 | Finish survey by June 2021
  Short Form Healthy Survey 36(SF-36) is used as a method of indirectly calculating the Health related quality of life from various aspects. The Short Form Healthy Survey 36(SF-36) consists of 36 questions (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health) that ask about the current state of health. In this study, SF-36v2™ Health Survey 1996, 2004 Health Assessment Lab, Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (IQOLA SF-36v2 Standard, Korea (Korean)) will be used
Patient Global Impression of Change (PGIC) | Finish survey by June 2021
  PGIC is an indicator that evaluates the improvement of patients in 5 steps, and the subject responds with improvement of functional limitation after treatment with 5 likert. (1=completely improved, 2=distinctly improved, 3=improved, 4=no significant difference, 5=worsened)
Spine surgery | Finish survey by June 2021
  The number of spinal surgery after treatment
Latest treatment | Finish survey by June 2021
  Latest treatment history about Failed Back Surgery Syndrome
Improvement of patients | Finish survey by June 2021
  5 steps (1=completely improved, 2=distinctly improved, 3=improved, 4=no significant difference, 5=worsened) are used to evaluate the improvement of patients
Patient satisfaction | Finish survey by June 2021
  7 steps (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse) are used to evaluate the satisfaction of patients
Return to daily life | Finish survey by June 2021
  How helpful treatment has been for returning to work and adjusting to daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province, South Korea

IPD SHARING:
Plan to Share IPD: No